CLINICAL TRIAL: NCT00838227
Title: Modafinil Augmentation in Chronic Schizophrenia and Schizoaffective Disorder: A Pilot Study
Brief Title: Modafinil Augmentation in Chronic Schizophrenia and Schizoaffective Disorder
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No source of funding to implement the study.
Sponsor: Manhattan Psychiatric Center (Other)
Responsible Party: Principal Investigator, Jean-Pierre Lindenmayer, Study Principal Investigator, Manhattan Psychiatric Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07I/C41-00
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Cognition; Obesity; Sedation
MeSH Terms: conditions — Schizophrenia; Obesity | interventions — Modafinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- One arm (Experimental): Study withdrawn due to lack of funds.
  Interventions: Drug: modafinil

INTERVENTIONS:
Drug: modafinil — Modafinil up to 400 mg daily will be added to a stable antipsychotic regimen
  Other Names: Provigil

SUMMARY:
This is an open label 8-week trial of modafinil up to 400 mg daily added to a stable antipsychotic regimen to evaluate the effect modafinil on cognition, sedation, and weight in patients with chronic schizophrenia. We hypothesize that modafinil, a wake-promoting agent, will lead to improved cognition, increased wakefulness, and decreased weight in patients with schizophrenia who are on stable antipsychotic regimens

DETAILED DESCRIPTION:
This study was withdrawn due to no source of funding to implement the study. No participants were enrolled for this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual-IV diagnosis of schizophrenia (all subtypes), illness duration greater than three years
* Auditory and visual acuity adequate to complete cognitive tests
* Stable dose of antipsychotics for at least 2 weeks prior to entry
* Good physical health determined by complete physical examination, laboratory tests, and EKG
* Capacity and willingness to give written informed consent.

Exclusion Criteria:

* Inability to read or speak English
* Documented disease of the central nervous system
* History of intellectual impairment pre-dating onset of symptoms of psychosis (e.g. mental retardation)
* Clinically significant or unstable cardiovascular, renal, hepatic, gastrointestinal, pulmonary or hematologic conditions;
* HIV positive
* Patients on antidepressants, including monoamine oxidase inhibitors
* Uncontrolled hypertension
* Pregnancy
* Patients with a current diagnosis of substance dependence
* Significant history of violence
* History of an eating disorder
* Ready for discharge within the following 8 weeks.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-02; Primary Completion 2012-01 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Cognitive changes as measured by the NIH MATRICS - Consensus Cognitive Battery (MCCB) | 8 weeks
  Study withdrawn due to lack of funds.

SECONDARY OUTCOMES:
Sedation and weight changes | 8 weeks
  Study withdrawn due to lack of funds.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Lindenmayer, MD, Principal Investigator — Manhattan Psychiatric Center

REFERENCES:
- [Background] Saavedra-Velez C, Yusim A, Anbarasan D, Lindenmayer JP. Modafinil as an adjunctive treatment of sedation, negative symptoms, and cognition in schizophrenia: a critical review. J Clin Psychiatry. 2009 Jan;70(1):104-12. doi: 10.4088/jcp.07r03982. Epub 2008 Nov 18. PMID 19026265